CLINICAL TRIAL: NCT00783783
Title: CYP2D6 PHARMACOGENETICS IN RISPERIDONE-TREATED CHILDREN AND ADOLESCENTS WITH PSYCHIATRIC OR NEURODEVELOPMENTAL DISORDERS
Brief Title: CYP2D6 Pharmacogenetics in Risperidone-Treated Children
Status: Completed | Type: Observational
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Ohio State University (Other); Rainbow Babies and Children's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2008-0659; SPR104683
Record Dates: First submitted 2008-10-31; First posted 2008-11-03 (Estimated); Last update posted 2012-12-11 (Estimated); Status verified 2012-12

CONDITIONS: Psychiatric Disorders; Neurodevelopmental Disorders
Keywords: Psychiatric disorders; Neurodevelopmental disorders; Autism; Risperidone; Pharmacogenetics; Pharmacokinetics
MeSH Terms: conditions — Mental Disorders; Neurodevelopmental Disorders; Autistic Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA from blood, buccal swab, or saliva
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Poor metabolizers: Patients with CYP2D6 genotypes predictive of poor metabolizer phenotype
- Non poor metabolizers: Patients with CYP2D6 genotypes predictive of intermediate, extensive, or ultra-rapid metabolizer phenotypes

SUMMARY:
Risperidone is an important medication used to treat children with psychiatric illnesses or neurodevelopmental disorders, such as autism. Despite excellent symptom control, the potential for side effects is worrisome. Treating these disorders is difficult because not everyone responds the same way to the same risperidone dose. One reason for this is genetic differences in how people break down the drug. Understanding these differences will help clinicians choose a dose and better predict the response so patients will be treated successfully with a lower risk for side effects. This study will research these genetic differences in children with psychiatric or neurodevelopmental disorders. Hypothesis: The inter-patient variability in risperidone pharmacokinetics and exposure, adverse events, and clinical response in patients with psychiatric or neurodevelopmental disorders is associated with identifiable pharmacogenetic factors, such as CYP2D6 single nucleotide polymorphisms (SNPs).

ELIGIBILITY:
Inclusion Criteria:

* Previous risperidone PK study participation (CCHMC, Rainbow Babies and Children's Hospital or OSU)
* CYP2D6 PM predicted phenotype
* Actively taking risperidone
* Under 18 years of age at time of enrollment
* Signed, dated informed consent forms

Exclusion Criteria:

* Investigators are unable to contact the subject/legal guardian(s)
* Subject is no longer taking risperidone
* CYP2D6 predicted phenotype other than PM
* Subject is non-White, with respect to race, for PK study participation
* Subject is 18 years of age or older
* Subject is less than 5 years of age
* Subject is pregnant at the time of the full PK study
* Subject/legal guardian unwilling or unable to participate in the study

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Subjects will include up to 41 risperidone-treated children and adolescents with psychiatric or neurodevelopmental (ND) disorders who participated in one of two previous risperidone pharmacokinetics investigations.
  To have a larger sample of poor metabolizer subjects, we plan to enroll at least 8 additional subjects who are on stable treatment with risperidone, and perform risperidone pharmacokinetics analyses. Prospectively enrolled subjects (n = 8) will be CYP2D6 poor metabolizers and will include White / Caucasian subjects, of any socioeconomic status, and will be recruited from inpatients or outpatients at Cincinnati Children's Hospital
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2008-11; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
association of common CYP2D6 polymorphisms with risperidone area under the curve | pre-dose (sample 1 = 0-30 minutes before first oral dose), and three at well-timed post-dose points (sample 2 = 15-30 minutes after dose; sample 3 = 60-90 minutes after dose; sample 4 = 4-6 hours after dose)

CONTACTS AND LOCATIONS:
Overall Officials: Shannon N Saldana, PharmD, MS, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

REFERENCES:
- [Background] Aman MG, Vinks AA, Remmerie B, Mannaert E, Ramadan Y, Masty J, Lindsay RL, Malone K. Plasma pharmacokinetic characteristics of risperidone and their relationship to saliva concentrations in children with psychiatric or neurodevelopmental disorders. Clin Ther. 2007 Jul;29(7):1476-86. doi: 10.1016/j.clinthera.2007.07.026. PMID 17825699
- [Background] Cabovska B, Cox SL, Vinks AA. Determination of risperidone and enantiomers of 9-hydroxyrisperidone in plasma by LC-MS/MS. J Chromatogr B Analyt Technol Biomed Life Sci. 2007 Jun 1;852(1-2):497-504. doi: 10.1016/j.jchromb.2007.02.007. Epub 2007 Feb 15. PMID 17344104
- [Result] Sherwin CM, Saldana SN, Bies RR, Aman MG, Vinks AA. Population pharmacokinetic modeling of risperidone and 9-hydroxyrisperidone to estimate CYP2D6 subpopulations in children and adolescents. Ther Drug Monit. 2012 Oct;34(5):535-44. doi: 10.1097/FTD.0b013e318261c240. PMID 22929407